CLINICAL TRIAL: NCT05698693
Title: Social Determinants of Sleep and Obesity: Culturally Informing a Sleep Extension Intervention for African American Adults
Brief Title: Social Determinants of Sleep and Obesity
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2022LS170
Record Dates: First submitted 2023-01-04; First posted 2023-01-26 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Insufficient Sleep; Physical Inactivity; Sedentary Behavior; Obesity
MeSH Terms: conditions — Sleep Deprivation; Sedentary Behavior; Obesity

STUDY DESIGN:
Intervention Model Description: The study uses qualitative interviews (Aim 1; n=10) to inform the adaptation of a sleep intervention for African American adults with overweight/obesity, short sleep, and physical inactivity. The feasibility, satisfaction, and preliminary efficacy will be tested (Aim 2) using a 2-armed randomized control trial (n=80).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep intervention (Experimental): The sleep extension intervention is a 4-week intervention consisting of weekly one-on-one contact with the goal of increasing total sleep time by 60 minutes by the end of four weeks conducted by Dr. Wu or a trained counselor. The first session will last 60 minutes and the content will include psychoeducation about the importance of sleep, sleep guidelines and target setting, and basic sleep hygiene. Participants in this condition will receive hardcopy weekly daily diary worksheets, and receive an online version of the sleep daily diary every morning to complete via text messaging. Sessions 2-4 will be between 15-30 minutes where Dr. Wu or a trained counselor will review the sleep diary, problem solve barriers to weekly goals, and sleep promoting behaviors will be reinforced. Material that would be covered during a missed session will be included in the next session the participant attends.
  Interventions: Behavioral: Sleep intervention
- Contact control (Active Comparator): The content of the contacts for this intervention condition will be based on the National Center for Healthy Housing's Healthy Homes program, a program designed by the UT School of Public Health. Participants in this condition will meet with Dr. Wu or a trained research staff member. They will meet through Zoom once a week for four sessions to go through each educational module. Sessions will conclude with the development of an action plan for participants. Staff will check in with participants regarding whether they were able to complete the tasks on their action plan, and if not, the reasons for this and potential strategies that may facilitate completion.
  Interventions: Behavioral: Contact Control

INTERVENTIONS:
Behavioral: Sleep intervention — The sleep extension intervention is a 4-week intervention consisting of weekly one-on-one contact with the goal of increasing total sleep time by 60 minutes by the end of four weeks conducted by Dr. Wu or a trained counselor.
  Arms: Sleep intervention
Behavioral: Contact Control — This is healthy homes intervention.The program provides education on healthy homes, provide advice on specific healthy homes problems, and recommend actions to be taken by families, landlords, and community members.
  Arms: Contact control

SUMMARY:
African American adults sleep less and obtain worse quality sleep compared to the national average, and emerging evidence links inadequate sleep with greater morbidity and mortality from chronic diseases such as diabetes, obesity, and cancer. To address this public health concern, the proposed research seeks to use a multi-method approach to adapt a sleep intervention for African American adults with overweight/obesity not meeting national sleep duration or physical activity recommendations. The overall goal of the project is to reduce cancer and obesity-related health disparities among African Americans.

ELIGIBILITY:
Inclusion Criteria:

* Not meeting Physical Activity Guidelines
* age range: 21 to 65 years
* body mass index range: 25.0 to 40 kg/m2
* average self-reported habitual sleep duration of ≤6 hours
* self-identify as Black or African American.

Exclusion Criteria:

* Self-reported organ-related disorder (COPD, cardiac arrhythmia, gastro-esophageal disorder)
* pregnant or less than 4 months postpartum
* infant living in household less than 1 year old

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility | 4 weeks
  Feasibility is achieved if intervention adherence is 75% across participants in the intervention group.
Satisfaction | 4 weeks post-intervention
  Satisfaction is achieved if the average score ≥20 on the Client Satisfaction Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Wu, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No